CLINICAL TRIAL: NCT04097977
Title: Networked-Based Recovery With User Involvement for Young People With Mental Illness: A Nonrandomized Clinical Trial
Brief Title: Networked-Based Recovery With User Involvement
Acronym: RENEW-S
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never funded
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRURegionZealand2
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Psychiatric Hospitalization
Keywords: User involvement; Patient-reported outcomes; Networked-based recovery
MeSH Terms: interventions — Rehabilitation; Educational Status

STUDY DESIGN:
Intervention Model Description: The project is designed as a non-randomized intervention study with a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: RENEW in a psychiatric ward (Experimental): Intervention The RENEW-S intervention consists of two key elements: collaborative networking and a youth group that will form the basis of real user involvement.
  Interventions: Other: An educational support model called RENEW (Rehabilitation for Empowerment, Natural Support, Education and Work) targeting young people with mental health difficulties.
- Conventional clinical practice in a psychiatric standard ward (No Intervention): The comparison group patients were admitted to a standard psychiatric ward that offered conventional care.

INTERVENTIONS:
Other: An educational support model called RENEW (Rehabilitation for Empowerment, Natural Support, Education and Work) targeting young people with mental health difficulties. — An educational support model called RENEW (Rehabilitation for Empowerment, Natural Support, Education and Work).
  Intervention The RENEW-S intervention consists of two key elements: collaborative networking and a youth group.
  Network meetings The RENEW-S network meetings is fundamental for this approach. First meeting between the young person and the facilitator is about what the young person can expect, and information about the principles and ideas behind RENEW-S. The RENEW-S process consists of 4 general phases: 1) a mapping process 2) the development of a team to support goal attainment 3) implementing the plans 4) preparation for exiting RENEW.
  Youth group The group is structured around the same agenda each time, starting with a presentation round, followed by an activity within the topic of the day, and finishing with sharing experiences of the activity in plenum. The young people can find inspiration regarding themes and exercises in the RENEW manual.
  Arms: Intervention: RENEW in a psychiatric ward

SUMMARY:
Introduction Over the past 20 years there has been an overall deterioration in the mental health of young people. An increasing number of young people are diagnosed with emotional disorders such as anxiety and depression. Overall, mental health problems represent the greatest health burden among adolescents. This means that many young people have difficulties in meeting demands, and challenges in education and employment. Thus, it is estimated that up to 60% dropout in education is due to mental health problems. Therefore, an educational, well-coordinated and early intervention is needed to support the young person's recovery process by activating the young person's social network.

Methods Study design The project is designed as a non-randomized intervention study with a control group. Comparative analyzes will be performed with pre- and post-assessments, as outlined in Figure 1. The study involves a regional hospital in mental health and five municipalities. The trial takes place from January 2020 to December 2022.

Intervention The RENEW-S intervention consists of two key elements: collaborative networking and a youth group that will form the basis of real user involvement.

Study population The participants are young adults aged 18 - 30 years with experiences as an inpatient.

Procedure for recruitment Questionnaires administered to the patients within the first 48 hours after admission, at discharge, 1 month after discharge and 3 months after discharge (Figure 1). Patients who did not consent to participation or failed to complete the questionnaire at the beginning of their stay were excluded from the study, as were those hospitalized for less than a week.

Ethics Information of participants and data management is in accordance with the Helsinki Declaration. The project is reported to the Danish Data Protection Agency and the Region Zealand Ethics Committee. Data are entered into the EasyTrial © Online Clinical Trial Management system. All personal identifiers will be removed or disguised during analysis to preclude personal identification.

DETAILED DESCRIPTION:
Introduction Over the past 20 years there has been an overall deterioration in the mental health of young people. An increasing number of young people are diagnosed with emotional disorders such as anxiety and depression. Overall, mental health problems represent the greatest health burden among adolescents. This means that many young people have difficulties in meeting demands, and challenges in education and employment. Thus, it is estimated that up to 60% dropout in education is due to mental health problems. Therefore, an educational, well-coordinated and early intervention is needed to support the young person's recovery process by activating the young person's social network.

In 1996, a group of US researchers and practitioners initiated an educational support model called RENEW (Rehabilitation for Empowerment, Natural Support, Education and Work) targeting young people with mental health difficulties. The primary goal of RENEW is to enhance young people's well-being through social inclusion and education, focusing on building young people's own capacities by supporting them in utilizing their existing social networks and adding new contacts in their path towards education and work. This support model has shown positive results with young people, where in particular their educational attainment and self-reported level of function have been improved. In 2013, the Psychiatric Center in Ballerup (Denmark) and the University of New Hampshire (USA) established a collaboration to investigate whether RENEW could be implemented in a Danish psychiatric setting, and achieve positive results as well. Young people with mental health difficulties have expressed lack of coherence in their pathways, which may result that the young people's problems are not dealt with in a timely manner, so that their problems worsen. It also means, there is a high risk that they will abandon education and become increasingly ill. New research by Tew et al also suggests that the network may have a greater impact than conventional treatment for young people with mental disorders. Thus, the Psychiatric Center in Ballerup wanted to create a greater degree of cohesion for the young people in their pathways across services through stronger cross-sectoral and team-based collaboration.

The Psychiatric Center Ballerup model has primarily focused on young outpatients and in municipal context. However, since the young inpatients usually have a greater need for support both in terms of their mental state, but also in relation to educational support and to support the young person's social network. Consequently, an improved intervention is needed to target this group: In order to prevent the development and aggravation of mental illness, there is a need for early intervention, recovery and inclusion of people with mental illness in education, work and everyday life. This project is based on the RENEW model and rooted in Psychiatry in Slagelse: RENEW-S. There is also a great desire for a high degree of user involvement in the project, partly for the purpose of learning for all parties involved, and partly to strengthen implementation. Involving users in the research project will enhance our understanding of young adults' perspectives in relation to the young person's hospitalization, social network, own resources and network based recovery. However, there is a lack of stakeholder involvement in this type of research. Co-operative inquiry is a research method that involves stakeholders such as service users and health professionals, as co-researchers. In co-operative inquiry, the production of knowledge is a joint venture among stakeholders and researchers who work together to create relevant and practice-oriented knowledge by means of the three following research steps: preparation, intervention and study outcomes assessment. The purpose of the project is to develop a network-based approach to the young inpatients with mental illness aged 18-30 years in order to strengthen the young person's social network and own resources using the RENEW model so that the young person achieves a higher degree of recovery, as well as education and employment.

Methods and analysis The research steps The research are involving the three steps: preparation, intervention and study outcomes assessment (see Table 1 for the timetable and tasks in relation to the research steps): A systematic review and focus interviews of young adults with mental illness together with health professionals are planned to inform the intervention. The preparation step regarding the systematic review is further explained in the Prospero protocol (ID: 151202). Likewise, further details concerning the planning and preparing of the focus group interviews are planned to be published as a study protocol in a qualitative journal.

Study design The project is designed as a non-randomized intervention study with a control group. Comparative analyzes will be performed with pre- and post-assessments, as outlined in Figure 1. The study involves a regional hospital in mental health and five municipalities. The trial takes place from January 2020 to December 2022.

Intervention The RENEW-S intervention consists of two key elements: collaborative networking and a youth group that will form the basis of real user involvement. The final version of the intervention can only be determined on the basis of the results of the research steps 1+2.

Network meetings The RENEW-S network meetings is fundamental for this approach. It is about using the young persons' network and their own available resources. The social network is of great importance to the young person's recovery process. First meeting between the young person and the facilitator is about what the young person can expect, and information about the principles and ideas behind RENEW-S. The RENEW-S process consists of 4 general phases: 1) a mapping process 2) the development of a team to support goal attainment 3) implementing the plans 4) preparation for exiting RENEW.

After finishing the mapping process, the young adults start working on their goals in collaboration with their support team, and participate in a weekly youth group (See Appendix: Additional description of the Network meetings).

Youth group The group is structured around the same agenda each time, starting with a presentation round, followed by an activity within the topic of the day, and finishing with sharing experiences of the activity in plenum. The young people can find inspiration regarding themes and exercises in the RENEW manual: Exercises include: 1) tasks and activities recommended by other young people or professionals 2) different recovery-oriented activities and cognitive / behavioral therapeutics exercises (25) 3) short films developed by the anti-stigma campaign "One of us" (2018) 4) field trips with a social purpose.

Training of facilitators and staff Facilitators are trained within each of the subject groups; nurse, doctor, physiotherapist, psychologist, and social worker. The training is planned to be conducted by the responsible project manager (RENEW) in Ballerup. The total staff will be introduced to the RENEW-S model at two initial workshops, as well as ongoing supervision every 14 days throughout the project period.

Setting The study took place at the Psychiatric Hospital in Slagelse, Denmark, which consists of four inpatient wards, an outpatient clinic, and an emergency ward serving a mixed urban and rural district. The department of psychiatry has 80 beds, 1995 discharges, and 39,391 visits to its outpatient clinics per year (2017 figures, obtained from HR department, Mental Health Services, Slagelse). As part of the publicly funded hospital services, the mental health services are administered by Region Zealand, one of Denmark's five regional health authorities, serving a population of 821,000.

Study population The participants are young adults aged 18 - 30 years with experiences as an inpatient. The study include inpatients admitted from October 2020 to April 2022, and the patients suffered from psychiatric disorders such as schizophrenia, psychosis, major depression, bipolar disorder, and severe personality disorder.

Procedure for recruitment Questionnaires administered to the patients within the first 48 hours after admission, at discharge, 1 month after discharge and 3 months after discharge (Figure 1). Patients who did not consent to participation or failed to complete the questionnaire at the beginning of their stay were excluded from the study, as were those hospitalized for less than a week.

Sample size The sample size calculation is based on an intervention study with SF-36 as the primary outcome, also conducted in Psychiatry (23). In this study, there is a clinically relevant effect size 0.5 with a power 80 ((α = 0.05). Based on this study's sample size calculation, 120 patients in each group are needed (intervention and control).

Data analysis Descriptive analysis Categorical data will be presented by numbers and proportions; continuous variables are shown by median and quartiles. Baseline data will be compared between the groups. The X2 test or Fisher's exact test are used for the analysis of categorical variables. For analysis of varians (ANOVA) and Kruskal -Wallis test are used for non-parametric and non-normally distributed variables, respectively.

Primary and secondary analysis All analyses will be conducted based on the intention-to-treat principle. Missing outcomes will be imputed and for non-adherence to protocol, a per-protocol analysis will be conducted as sensitivity analysis. A non-response analysis will be carried out for excluded patients and non-completers.

Ethics and dissemination Information of participants and data management is in accordance with the Helsinki Declaration. The project is reported to the Danish Data Protection Agency and the Region Zealand Ethics Committee. Data are entered into the EasyTrial © Online Clinical Trial Management system. All personal identifiers will be removed or disguised during analysis to preclude personal identification. The following articles are planned for publication: 1) The effects of networked based recovery in a mental health setting: findings from a systematic review 2) Networked-based recovery in mental health: Inpatient experiences 3) Improved patient-reported outcomes after network-based recovery to young adults in mental health: A nonrandomized clinical trial

Organization The project is organized with a steering group, a project group. All groups include users with experiences from hospitalization in mental health services, health professionals and researchers. The steering group is responsible for the project being implemented in accordance with the project description, deciding on changes and approving the framework and resources. The steering group consists of two users, who have been hospitalized and diagnosed with a psychiatric diagnoses, and involved in other projects with user involvement. The project group is responsible for day-to-day operations, including ensuring that the project's stakeholders are involved in the process, as well as conducting the actual intervention, such as assessments of impact, and application for external funds. Moreover, recruitment of project staff and information about the project. The project group is also responsible for ensuring the necessary research strength in the study design, methods and analyses, including publication of results. The project group consists of five users from the user panel in Psychiatry in Region Zealand.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 18 - 30 years
* Diagnosed with a mental disorder
* Have experienced hospitalization

Exclusion Criteria:

* Cognitive deficit
* Patients who did not consent to participation
* Hospitalized for less than a week

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mental health status. | At baseline and after 4 months.
  Mental health status is valid and reliable indicator of the patients self-reported mentale state and well-being. Mental status is assessed using the standardized Short Form Health Survey (SF-36). Scores range from 0 (zero) to 100, with higher scores indicating better health.

SECONDARY OUTCOMES:
Change in Level of function. | At baseline and after 4 months.
  The young adults' level of function is assessed using the Global assessment of functioning (GAF). Scores range from 0 to 100, with higher scores indicating better health.
Change in Patient satisfaction. | At baseline and after 4 months.
  Satisfaction is measured with the client satisfaction score scale (CSQ-8). Total scores range from 8 to 32, with higher scores indicating greater satisfaction.
Change in Recovery. | At baseline and after 4 months.
  The patients' recovery will be assessed by the 24-item recovery assessment scale-revised (RAS-R). Score range of 46-120, with higher scores indicating a higher degree of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marcussen, Dr., Principal Investigator — University of Southern Denmark, Denmark.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGorry PD. The specialist youth mental health model: strengthening the weakest link in the public mental health system. Med J Aust. 2007 Oct 1;187(S7):S53-6. doi: 10.5694/j.1326-5377.2007.tb01338.x. PMID 17908028
- [Background] Andreasen J, Poulsen S, Hoej M, Arnfred S. 'It is important for us to see the mentors as persons' - participant experiences of a rehabilitation group. Int J Qual Stud Health Well-being. 2019 Dec;14(1):1632108. doi: 10.1080/17482631.2019.1632108. PMID 31238817
- [Background] Hunt J, Eisenberg D. Mental health problems and help-seeking behavior among college students. J Adolesc Health. 2010 Jan;46(1):3-10. doi: 10.1016/j.jadohealth.2009.08.008. Epub 2009 Oct 20. PMID 20123251
- [Background] Waldemar AK, Esbensen BA, Korsbek L, Petersen L, Arnfred S. Recovery-oriented practice: Participant observations of the interactions between patients and health professionals in mental health inpatient settings. Int J Ment Health Nurs. 2019 Feb;28(1):318-329. doi: 10.1111/inm.12537. Epub 2018 Aug 27. PMID 30151987
- [Background] Buus N, Juel A, Haskelberg H, Frandsen H, Larsen JLS, River J, Andreasson K, Nordentoft M, Davenport T, Erlangsen A. User Involvement in Developing the MYPLAN Mobile Phone Safety Plan App for People in Suicidal Crisis: Case Study. JMIR Ment Health. 2019 Apr 16;6(4):e11965. doi: 10.2196/11965. PMID 30990456
- [Background] Berring LL, Hummelvoll JK, Pedersen L, Buus N. A Co-operative Inquiry Into Generating, Describing, and Transforming Knowledge About De-escalation Practices in Mental Health Settings. Issues Ment Health Nurs. 2016 Jul;37(7):451-63. doi: 10.3109/01612840.2016.1154628. Epub 2016 Apr 12. PMID 27070499
- [Background] Hendryx M, Green CA, Perrin NA. Social support, activities, and recovery from serious mental illness: STARS study findings. J Behav Health Serv Res. 2009 Jul;36(3):320-9. doi: 10.1007/s11414-008-9151-1. Epub 2008 Nov 15. PMID 19011972
- [Background] Richards DA, Bower P, Chew-Graham C, Gask L, Lovell K, Cape J, Pilling S, Araya R, Kessler D, Barkham M, Bland JM, Gilbody S, Green C, Lewis G, Manning C, Kontopantelis E, Hill JJ, Hughes-Morley A, Russell A. Clinical effectiveness and cost-effectiveness of collaborative care for depression in UK primary care (CADET): a cluster randomised controlled trial. Health Technol Assess. 2016 Feb;20(14):1-192. doi: 10.3310/hta20140. PMID 26910256
- [Background] Andriessen K. Suicide bereavement and postvention in major suicidology journals: lessons learned for the future of postvention. Crisis. 2014;35(5):338-48. doi: 10.1027/0227-5910/a000269. PMID 25163845
- [Result] Patel V, Flisher AJ, Hetrick S, McGorry P. Mental health of young people: a global public-health challenge. Lancet. 2007 Apr 14;369(9569):1302-1313. doi: 10.1016/S0140-6736(07)60368-7. PMID 17434406